CLINICAL TRIAL: NCT01372046
Title: Implementing & Testing Assessment and Referral Technologies in Juvenile Justice
Acronym: JAARP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: George Mason University (Other)
Collaborators: University of Maryland (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Faye S Taxman, Ph.D., Univeristy Professor, George Mason University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA018759 (NIH); R01DA018759 (NIH)
Record Dates: First submitted 2011-06-10; First posted 2011-06-13 (Estimated); Last update posted 2011-06-13 (Estimated); Status verified 2009-06

CONDITIONS: Skill Development of Staff; Use of Standardized Assessment Tools
Keywords: technology transfer; skill development; organizational change

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Enhanced (Experimental): A external consultant works with the team to develop skills and trains an in-house coach
  Interventions: Behavioral: Booster Sessions
- Trainer (Experimental): External consultant provides booster session
  Interventions: Behavioral: Booster Sessions
- Standard (Experimental): Receive agency training
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Booster Sessions — Provides onsite booster sessions for one year to the group after participating in standard care
  Arms: Enhanced; Trainer
Behavioral: Training — memorandums, staff meetings
  Arms: Standard

SUMMARY:
1. Assess the impacts of implementing a juvenile assessment, referral, placement, and treatment planning (J-ARPP) protocol, and of different strategies for transferring J-ARPP technology, on service utilization of youth entering the juvenile justice system.
2. Assess the impacts of implementing J-ARPP, and of different strategies for transferring J-ARPP technology, on measures of organizational readiness and motivation, and staff attitudes about assessment and service.
3. Assess the impacts of implementing J-ARPP, and of different strategies for transferring J-ARPP technology, on measures of systems integration.
4. Assess fidelity to the J-ARPP protocol and the relationship between fidelity to the J-ARPP protocol and service utilization of youth entering the juvenile justice system.

ELIGIBILITY:
Inclusion Criteria:

* all offices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Service utilization | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Faye Taxman, Ph.D., Principal Investigator — George Mason University; Doug Young, MA, Principal Investigator — University of Maryland
Locations (1):
- State of MD, Juvenile justice offices, Baltimore, Maryland, United States